CLINICAL TRIAL: NCT00266539
Title: Comparison of the Safety and Efficacy of Patient Controlled Analgesia Delivered by Fentanyl HCl Transdermal System Versus Morphine IV Pump for Pain Management After Non-emergent Abdominal or Pelvic Surgery
Brief Title: A Comparison of the Safety and Effectiveness of Two Forms of Patient-controlled Pain Medication Used After Scheduled Abdominal or Pelvic Surgery: The Fentanyl Transdermal System Versus the Morphine Intravenous Pump
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004717
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; patient-controlled analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

INTERVENTIONS:
Drug: E-TRANS Fentanyl hydrochloride; Morphine

SUMMARY:
The purpose of this study is to compare two pain medications delivered by two different forms of patient-controlled pain management systems: the Fentanyl HCl Patient-Controlled Transdermal System (E-TRANS fentanyl) and the morphine intravenous pump. Fentanyl HCl and morphine are narcotic pain relievers. The E-TRANS fentanyl system is a small unit worn on the patient's upper outer arm or chest that uses low-intensity electrical current to deliver fentanyl through the skin and into the patient's bloodstream. The patients studied will be those who have just had scheduled abdominal or pelvic surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare two pain medications delivered by two different forms of patient-controlled analgesia (PCA). PCA is a form of pain management that allows the patient to control the amount of pain medication he or she receives. The PCA E-TRANS fentanyl system is a credit card-sized unit that is worn on the patient's upper outer arm or chest. It uses low-intensity electrical current to move fentanyl through the skin and into the patient's bloodstream. It does not require the insertion of an intravenous (IV) needle, or injection for pain management. PCA IV morphine is delivered into a vein by an IV infusion pump that is specially designed to be controlled by the patient. The PCA E-TRANS fentanyl system delivers a 40 microgram dose of fentanyl and the PCA IV morphine delivers a 1 milligram intravenous dose of morphine. The patients in this study are those scheduled for non-emergent abdominal or pelvic surgery. Before surgery, patients will be taught how to use both PCA devices, and randomly assigned to receive either PCA IV morphine or E-TRANS fentanyl. After undergoing surgery, patients will have the PCA device applied to the skin (E-TRANS fentanyl) or an IV inserted into a vein (PCA IV morphine), according to the random assignment. The patient will then be allowed to control delivery of the assigned medication for 72 hours. During the first 24 hours, the patient will be asked about the amount of pain he or she is having. The primary measure of effectiveness is successful pain relief (defined by a rating of "Excellent", or "Good") on the 24-hour patient global assessment of the method of pain control. At 24, 48, and 72 hours, the patient will be asked a set of specific questions to measure the effectiveness of the PCA. In addition, the patient's doctor, and nurses, will answer questions about the PCA system. Safety will be assessed by monitoring the patient's vital signs and recording any adverse events, including problems at the location on the patient's body where the PCA device has been applied or inserted. The objective is to establish that the Fentanyl HCl Patient-Controlled Transdermal System (E-TRANS fentanyl) is as effective as intravenous (IV) PCA morphine in controlling pain after non-emergent abdominal or pelvic surgery.

E-TRANS fentanyl 40 mcg transdermally per patient-activated dose over 10 minutes, up to 6 doses per hour or a maximum of 80 doses in 24 hours; Patient controlled intravenous morphine 1 mg dose, up to 10 doses per hour or a maximum of 240 doses in 24 hours. Study duration is 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pre-operative American Society of Anesthesiology Physical Status I, II, or III (Class I are healthy persons less than 80 years of age, Class II are patients over age 80 years of age with mild systemic disease, and Class III are patients with severe and non-incapacitating disease)
* Admitted to the Post-Anesthesia Care Unit after general anesthesia or spinal/epidural anesthesia using short-acting agents
* Having had one of these surgical procedures: small and large bowel resections with anastomosis, colectomy, enterolysis, sigmoidectomy, closure of enteric fistulae, repair of cecal or sigmoid volvulus, lower anterior resection, stoma closure, bariatric surgery, liver resection, splenectomy, gastrectomy, fundoplication, total abdominal hysterectomy, total vaginal hysterectomy, anterior-posterior repair, oophorectomy, or myomectomy and cystectomy
* Awake and breathing spontaneously with a respiratory rate of 8 to 24 breaths per minute and oxygen saturation of 90% or higher (with or without supplemental oxygen)
* Expected to remain hospitalized for at least 24 hours postoperatively

Exclusion Criteria:

* Patients whose postoperative pain would normally be managed with oral or non-narcotic pain medication
* Who received long-acting intraoperative epidural, spinal anesthesia, or local anesthetics in the surgical area, or who are expected to have postoperative analgesia supplied by a continuous regional technique or patient-controlled epidural analgesia
* Have a history of allergy, hypersensitivity, or tolerance to fentanyl or morphine, have a history of allergy or hypersensitivity to cetylpyridinium chloride or skin adhesives, or have the presence of active skin disease that would interfere with application of the E-TRANS fentanyl system
* Who received steroids within 1 month before surgery or during surgery
* Expected to require intensive care postoperatively or who will probably need additional surgical procedures within 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2004-04; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Success (defined by a rating of "Excellent" or "Good") at the 24-hour patient global assessment of the method of pain control.

SECONDARY OUTCOMES:
Proportion of successes at 48 and 72 hours and at final assessment; mean pain intensity assessment at 24, 48, and 72 hours and at final assessment; mean scores from the Ramsay Sedation Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- [Result] Minkowitz HS, Rathmell JP, Vallow S, Gargiulo K, Damaraju CV, Hewitt DJ. Efficacy and safety of the fentanyl iontophoretic transdermal system (ITS) and intravenous patient-controlled analgesia (IV PCA) with morphine for pain management following abdominal or pelvic surgery. Pain Med. 2007 Nov-Dec;8(8):657-68. doi: 10.1111/j.1526-4637.2006.00257.x. PMID 18028044
- See also: Comparison of the Safety and Efficacy of Patient Controlled Analgesia Delivered by Fentanyl HCl Transdermal System Versus Morphine IV Pump for Pain Management after Non-emergent Lower Abdominal or Pelvic Surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=93&filename=CR004717_CSR.pdf